CLINICAL TRIAL: NCT03798223
Title: Optimal Treatment Protocol for Selective Laser Trabeculoplasty
Acronym: OSLT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Optimal SLT; 254861 (Other: FoU i VGR ID nr)
Record Dates: First submitted 2019-01-03; First posted 2019-01-09 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Glaucoma, Open-Angle; Pseudoexfoliation Glaucoma; Ocular Hypertension
Keywords: Selective Laser Trabeculoplasty
MeSH Terms: conditions — Glaucoma, Open-Angle; Exfoliation Syndrome; Ocular Hypertension

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The treatment protocol is masked for the patient and for the nurses conducting measures of intraocular pressure during follow-up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- 180/low (Experimental): SLT treatment in the lower half of the trabecular meshwork (180 degrees) consisting of 50+/-5 adjacent laser effects. The energy is adjusted 0,1 mJ below the threshold of formation of micro bubbles.
  Interventions: Procedure: SLT
- 180/high (Experimental): SLT treatment in the lower half of the trabecular meshwork (180 degrees) consisting of 50+/-5 adjacent laser effects. The energy is adjusted to achieve the formation of micro bubbles at 50-75% of laser effects.
  Interventions: Procedure: SLT
- 360/low (Experimental): SLT treatment in the full circumference of the trabecular meshwork (360 degrees) consisting of 100+/-10 adjacent laser effects. The energy is adjusted 0,1 mJ below the threshold of formation of micro bubbles.
  Interventions: Procedure: SLT
- 360/high (Experimental): SLT treatment in the full circumference of the trabecular meshwork (360 degrees) consisting of 100+/-10 adjacent laser effects. The energy is adjusted to achieve the formation of micro bubbles at 50-75% of laser effects.
  Interventions: Procedure: SLT

INTERVENTIONS:
Procedure: SLT — A drop of Pilocarpine 4% is administered to the eye 20 minutes before SLT. Immediately before SLT a drop of Tetracaine hydrochloride 1% is administered. Selective laser trabeculoplasty is conducted through a Latina lens, in a fashion determined by randomization to a study arm (see description).

SUMMARY:
A randomized controlled trial to evaluate which treatment protocol in selective laser trabeculoplasty that is most optimal in terms of efficacy and safety.

DETAILED DESCRIPTION:
A randomized controlled trial in which individuals scheduled for SLT are randomized to one of four treatment protocols, which represent the most common variants of the treatment in clinical use.

Treatment is performed either at 360 degrees or 180 degrees and with a laser energy level either 0,1 millijoules (mJ) below the microbubble formation limit ("low" energy) or at a level that gives microbubbles at 50-75% of laser effects ("high" energy). This gives four treatment arms: 180/low, 180/high, 360/low and 360/high. Group allocation is masked for the patient and is coded in the records.

The results for short and long term treatment effects are compared between the groups, as well as the complication rate and postoperative discomfort.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis primary open-angle glaucoma, pseudo-exfoliative glaucoma or ocular hypertension.
* intra-ocular pressure (IOP) at least 18 mmHg treatment day.
* treatment is performed by an experienced laser surgeon.
* SLT treatment and follow-up are expected to be possible to perform in an adequate way, considering anatomical factors, age and the general health of the patient.

Exclusion Criteria:

* change of IOP-lowering medication during the last three months.
* planned change of intra-ocular-pressure-lowering medication.
* previous glaucoma surgery (other than SLT and ALT)
* previous intra-ocular surgery during the last three months.
* previous intra-ocular inflammatory disease during the last year.
* planned intra-ocular surgery.
* hyper-pigmented anterior chamber angle.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in intraocular pressure (IOP) | Before SLT and thereafter regularly for 3 years
  The IOP is measured with a Goldmann Applanation Tonometer (GAT) three times before SLT and then at regular intervals after the procedure. The reduction is registered and analyzed in absolute (mmHg) and relative (percent of the IOP before SLT) measures.
  Measurement of IOP is planned 1, 3, 6 and 12 months post SLT, and thereafter every six months for 3 years after SLT. The study is conducted in a regular clinical setting and the above mentioned times might be delayed. If target pressure is not achieved, measurements will be planned at shorter intervals, according to a specified algorithm, due to safety reasons.
Achievement of 20% reduction in IOP | For 3 years
  See Outcome 1. Analysis of differences between the study arms will also be conducted measuring the proportion of eyes achieving 20% reduction in IOP or more at different time points in each group.
Survival (no additional intervention) | For 3 years
  Kaplan-Meier survival analysis will be conducted, measuring the proportion of eyes that stay in the study groups but do not receive any further IOP-lowering intervention (medical, surgical or laser).

SECONDARY OUTCOMES:
Survival (SLT allowed) | For 3 years
  See Outcome 3. Kaplan-Meier survival analysis is performed the same way, but additional SLT-treatment will not be judged as failure.
Pain perioperatively: on a scale | Immediately after treatment
  The patient will grade perioperative pain on an arbitrary scale between 0 (no pain) and 4 (maximum pain) on a written protocol.
Pain postoperatively: on a scale | During the first month
  The patient will grade post-operative pain on an arbitrary scale between 0 (no pain) and 4 (maximum pain) on a written protocol, also stating the duration of pain.
Light sensitivity postoperatively | During the first month
  The patient will grade post-operative sensitivity to light on an arbitrary scale between 0 (no difference) and 4 (very intense sensitivity to light) on a written protocol, also stating the duration of light sensitivity.
Impairment of vision postoperatively | During the first month
  The patient will grade post-operative impairment of vision on an arbitrary scale between 0 (no difference) and 4 (cannot see ones own hand) on a written protocol, also stating the duration of vision impairment.
Redness postoperatively | During the first month
  The patient will grade post-operative redness of the eye on an arbitrary scale between 0 (no difference) and 4 (very intense redness) on a written protocol, also stating the duration of redness.
Flare (inflammation measurement of the anterior chamber) | Pre-operatively and then one day, one week and one month post-operatively.
  15 participants from each treatment arm (60 in total, randomized in a separate block after informed consent) will undergo measurement with a Laser Flare Meter.
Adverse events | 3 years (although adverse events, if any, are anticipated to emerge in the first post-operative days or weeks).
  The type and frequency of adverse events will be recorded and analyzed in each of the study arms.

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo Ayala, MD, PhD, Study Chair — Vastra Gotaland Region; Tobias Dahlgren, MD, Principal Investigator — Vastra Gotaland Region
Locations (4):
- Sweden (4):
  - Ogonkliniken, Sodra Alvsborgs Sjukhus, Borås, Västra Götaland County
  - Ogonkliniken, Sahlgrenska Universitetssjukhuset, Mölndal, Västra Götaland County
  - Ogonkliniken, Skaraborgs Sjukhus, Skövde, Västra Götaland County
  - Ogonkliniken NU-sjukvarden, Uddevalla, Västra Götaland County

IPD SHARING:
Plan to Share IPD: No